CLINICAL TRIAL: NCT06738095
Title: Effect of Low-level Red-light on Ultra-high Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, cao kai, Dr, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingTH TRECKY239
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2022-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- red-light (Experimental): Children with ultra-high myopia were treated with daily low-level red-light, which was used twice a day, with four hours interval. Three minutes for each session of treatment
  Interventions: Device: daily low-level red-light

INTERVENTIONS:
Device: daily low-level red-light — Daily low-level red-light is a kind of myopia intervention. Red-light typically using 650-nm wave of length. The treatment duration last 3 minutes each time, every day children were anticipated to use two times, at home.

SUMMARY:
100 eyes of ultra-high myopia were treated with daily low-level red-light. The age of children ranged from 3 to 16.3 years. The follow-up duration was one year. The objective was to explore the effect of daily low-level red-light on ultra-high myopia treatment

ELIGIBILITY:
Inclusion Criteria:

A. The age is over 3 years old and under 18 years old. B. The spherical equivalent error is ≤ -6 D diopter . D. be able to cooperate to complete various eye examinations. E. be able to attend follow-up according to the specified time. F the guardian can accompany the use of the instrument.

Exclusion Criteria:

A. Complications associated with high myopia (such as choroidal neovascularization, macular split or hole, Rhegmatogenous retinal detachment); B other macular diseases (central serous retinopathy) or other eye diseases (e.g.Glaucoma, cataract, uveitis); C complicated with photosensitivity, psoriasis, albinism, hyperactivity disorder, nephrotic syndrome and systemic erythema Immune system diseases such as lupus; D. other systemic diseases or pregnancy; E. other similar instruments have been used for treatment in the past six months.

F. can't cooperate to complete various eye examinations. G. The guardian cannot accompany the use of this instrument.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Changes in axial length | one year
  One year changes in axial length

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided